CLINICAL TRIAL: NCT06113835
Title: Viable Myocardium Detected by the Combination of Hybrid PET/MR and SPECT Imaging for the Prediction of the Efficacy of PCI in Patients With Chronic Total Occlusion.
Brief Title: Viable Myocardium Detected by Hybrid PET/MR and SPECT for the Prediction of the Efficacy of PCI in Patients With CTO.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Director of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 022
Record Dates: First submitted 2023-10-30; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: Chronic Total Occlusion of Coronary Artery; viable myocardium; Hybrid PET/MR and SPECT Imaging; Percutaneous coronary intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- successful group: CTO PCI Technical success ,deployment of a balloon or stent with final antegrade TIMI flow grade 2 or 3, residual stenosis <30% , and no significant side branch occlusion.
  Interventions: Procedure: CTO PCI
- unsuccessful group: CTO PCI Technical unsuccess
  Interventions: Procedure: CTO PCI

INTERVENTIONS:
Procedure: CTO PCI — percutaneous coronary intervention

SUMMARY:
CTO intervention is controversial, and viable myocardium is critical to the improvement of cardiac function and prognosis of patients. However, it remains uncertain whether viable myocardium detected by Hybrid PET/MR and SPECT Imaging improves the PCI efficacy in Patients With CTO.

In this investigator-initiated, prospective, single-center, observational trial, patients meeting the inclusion/exclusion criteria would be assigned to the successful group or the unsuccessful group based on the success of PCI, both undergoing pre-operative and 6-month follow-up Hybrid PET/MR and SPECT imaging. The improvement of left ventricular (LV) recovery after 6 months will be observed.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) for chronic total occlusion (CTO) represents a major challenge in interventional cardiology. However, the results of the current large-scale CTO study showed that PCI failed to improve the long-term prognosis (MACE) over medical therapy. Is CTO intervention necessary and how to select appropriate patients for intervention? Previous studies have found the presence and improvement of viable myocardium(VM) in patients with CTO after PCI，and the amount of preoperative VM is critical to the choice of treatment for patients.

Several diagnostic techniques have been introduced to assess myocardial viability and LV recovery, allowing the identification of ischemic myocardium with potentially reversible systolic dysfunction, such as hibernating myocardium, among which 2-deoxy-2-[18F]fluoro-D-glucose positron emission tomography ( 18F-FDG PET) as the "gold standard" for clinical assessment of VM. However, single FDG-PET assessment of VM has limitations and cannot accurately identify hibernating myocardium. 99mTc-Methoxyisobutylisocyanide single-photon emission computed tomography (99mTc-MIBI SPECT), as a validated method for assessing myocardial perfusion, is recommended by guidelines for the assessment of VM in combination with FDG-PET. In recent years, contrast-enhanced cardiac magnetic resonance imaging (cardiac magnetic resonance imaging CMR) has been increasingly used to assess myocardial viability due to its high spatial resolution, which allows the acquisition of cardiac function and myocardial scarring.

However, there are fundamental differences between the two methods in assessing VM and LV function, with LGE-CMR primarily describing an increase in extracellular space associated with scar tissue, whereas FDG-PET uptake represents the true metabolic signals of viable cardiomyocytes. They are complementary.

Hybrid PET/MRI has recently been used as a novel modality for evaluating cardiac diseases, allowing a truly synchronous/simultaneous acquisition of complementary information such as high-resolution anatomy and myocardial metabolism in merged images. However, few studies about PET/MRI were done in patients with CTO.

Our study aims to investigate the effect of CTO-PCI by assessing VM detected by the combination of PET/MR and SPECT and to investigate the predictive value of viable myocardial area on the efficacy of CTO-PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≧ 18 years, < 75 years;
2. complete occlusion of the coronary artery, confirmed by coronary angiography with TIMI flow grade 0, and occlusion for ≥3 months;
3. presence of angina or angina-equivalent symptoms ; undergo coronary intervention;

Exclusion Criteria:

1. life expectancy < 1 year due to non-cardiac disease;
2. contraindications to SPECT/PET/MRI: pregnancy, contrast allergy, claustrophobia, history of pacemaker and ICD implantation, other ferromagnetic materials in the body;
3. acute coronary syndrome within the last 3 months;
4. severe valvular heart disease;
5. haemodynamic instability;
6. hepatic or renal insufficiency, with alanine aminotransferase (ALT) > 3 times the upper limit of normal or glomerular filtration rate ≤ 30 mL/min;
7. two or more CTO lesions;
8. previous myocardial infarction.
9. Others who, in the opinion o f the investigator, should not be enrolled;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with symptomatic coronary artery disease (CAD) (angina or angina equivalent) in the presence of a CTO of a relevant coronary artery
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
left ventricular ejection fraction increased by ≥5% | 6±1 month
  PET/MR postoperative follow-up
Segmental ventricular wall motion score decreased by ≥1 | 6±1 month
  PET/MR postoperative follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, Dr,PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azzalini L, Jolicoeur EM, Pighi M, Millan X, Picard F, Tadros VX, Fortier A, L'Allier PL, Ly HQ. Epidemiology, Management Strategies, and Outcomes of Patients With Chronic Total Coronary Occlusion. Am J Cardiol. 2016 Oct 15;118(8):1128-1135. doi: 10.1016/j.amjcard.2016.07.023. Epub 2016 Jul 28. PMID 27561190
- [Background] Hamzaraj K, Kammerlander A, Gyongyosi M, Frey B, Distelmaier K, Graf S. Patient Selection and Clinical Indication for Chronic Total Occlusion Revascularization-A Workflow Focusing on Non-Invasive Cardiac Imaging. Life (Basel). 2022 Dec 20;13(1):4. doi: 10.3390/life13010004. PMID 36675954
- [Background] Mehran R, Claessen BE, Godino C, Dangas GD, Obunai K, Kanwal S, Carlino M, Henriques JP, Di Mario C, Kim YH, Park SJ, Stone GW, Leon MB, Moses JW, Colombo A; Multinational Chronic Total Occlusion Registry. Long-term outcome of percutaneous coronary intervention for chronic total occlusions. JACC Cardiovasc Interv. 2011 Sep;4(9):952-61. doi: 10.1016/j.jcin.2011.03.021. PMID 21939934
- [Background] Henriques JP, Hoebers LP, Ramunddal T, Laanmets P, Eriksen E, Bax M, Ioanes D, Suttorp MJ, Strauss BH, Barbato E, Nijveldt R, van Rossum AC, Marques KM, Elias J, van Dongen IM, Claessen BE, Tijssen JG, van der Schaaf RJ; EXPLORE Trial Investigators. Percutaneous Intervention for Concurrent Chronic Total Occlusions in Patients With STEMI: The EXPLORE Trial. J Am Coll Cardiol. 2016 Oct 11;68(15):1622-1632. doi: 10.1016/j.jacc.2016.07.744. PMID 27712774
- [Background] Ryan M, Morgan H, Chiribiri A, Nagel E, Cleland J, Perera D. Myocardial viability testing: all STICHed up, or about to be REVIVED? Eur Heart J. 2022 Jan 13;43(2):118-126. doi: 10.1093/eurheartj/ehab729. PMID 34791132
- [Background] Ling LF, Marwick TH, Flores DR, Jaber WA, Brunken RC, Cerqueira MD, Hachamovitch R. Identification of therapeutic benefit from revascularization in patients with left ventricular systolic dysfunction: inducible ischemia versus hibernating myocardium. Circ Cardiovasc Imaging. 2013 May 1;6(3):363-72. doi: 10.1161/CIRCIMAGING.112.000138. Epub 2013 Apr 17. PMID 23595888
- [Background] Allman KC. Noninvasive assessment myocardial viability: current status and future directions. J Nucl Cardiol. 2013 Aug;20(4):618-37; quiz 638-9. doi: 10.1007/s12350-013-9737-8. Epub 2013 Jun 15. PMID 23771636
- [Background] Dilsizian V, Bacharach SL, Beanlands RS, Bergmann SR, Delbeke D, Dorbala S, Gropler RJ, Knuuti J, Schelbert HR, Travin MI. ASNC imaging guidelines/SNMMI procedure standard for positron emission tomography (PET) nuclear cardiology procedures. J Nucl Cardiol. 2016 Oct;23(5):1187-1226. doi: 10.1007/s12350-016-0522-3. Epub 2016 Jul 8. No abstract available. PMID 27392702
- [Background] Kwong RY, Chan AK, Brown KA, Chan CW, Reynolds HG, Tsang S, Davis RB. Impact of unrecognized myocardial scar detected by cardiac magnetic resonance imaging on event-free survival in patients presenting with signs or symptoms of coronary artery disease. Circulation. 2006 Jun 13;113(23):2733-43. doi: 10.1161/CIRCULATIONAHA.105.570648. Epub 2006 Jun 5. PMID 16754804
- [Background] Vitadello T, Kunze KP, Nekolla SG, Langwieser N, Bradaric C, Weis F, Cassese S, Fusaro M, Hapfelmeier A, Lewalter T, Schwaiger M, Kastrati A, Laugwitz KL, Rischpler C, Ibrahim T. Hybrid PET/MR imaging for the prediction of left ventricular recovery after percutaneous revascularisation of coronary chronic total occlusions. Eur J Nucl Med Mol Imaging. 2020 Dec;47(13):3074-3083. doi: 10.1007/s00259-020-04877-w. Epub 2020 May 30. PMID 32472438